CLINICAL TRIAL: NCT00520585
Title: Study of Influence of Atorvastatin on the Repolarisation Phase of Cardiomyocytes
Acronym: ATORVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Masaryk University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CS-15-11-2006
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Last update posted 2007-08-24 (Estimated); Status verified 2007-08

CONDITIONS: Heterogeneity of Cardiomyocytes Repolarisation; Autonomic Changes of Cardiomyocytes Repolarisation
Keywords: atorvastatin; repolarisation; cardiomyocytes
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: atorvastatin — atorvastatin 20 mg once vs. atorvastatin 80 mg once vs. placebo

SUMMARY:
The aim of this study is to evaluate influence of atorvastin on the repolarisation phase of cardiomyocytes. If there is any, it could be a part of positive "non-lipid" effect of statins in therapy of ischaemic heart disease.

Study hypothesis: atorvastin will decrease heterogeneity of repolarisation of cardiomyocytes in comparison with placebo

DETAILED DESCRIPTION:
The group will consist of 40 healthy volunteers. The study will be mono-centric. The repolarisation phase of cardiomyocytes will be evaluated using long - term 12-lead digital ECG monitoring. There will be 3 single ECG recordings - randomly after 20 mg of atorvastin, 80 mg of atorvastatin and placebo, respectively.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* age 18 - 45 years

Exclusion Criteria:

* no chronic active disease
* no concomitant pharmacotherapy, excluding hormonal contraception
* abnormal ECG, echocardiography, laboratory findings
* known hypersensitivity or myopathy due o statin
* pregnancy, lactation, breast implants
* skin disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-08; Study Completion 2007-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ondrej Toman, MD, Principal Investigator — University Hospital Brno, Department of Cardiology, Brno, Czech Republic